CLINICAL TRIAL: NCT01379365
Title: Cryo-Touch III Refinement Study Investigational Plan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-4500; MS-4500
Record Dates: First submitted 2011-06-20; First posted 2011-06-23 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Facial Wrinkles; Skin Aging
Keywords: wrinkle rhytid aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: Cryo-Touch III

INTERVENTIONS:
Device: Cryo-Touch III — Percutaneous treatment with the device

SUMMARY:
This is a prospective, non-randomized study to evaluate the performance of the MyoScience Cryo-Touch III device for the treatment of glabellar and/or forehead wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-70 years
* Subject has a glabellar and/or forehead wrinkle rating by investigator of at least 2 in animation on the 5-point Wrinkle Scale (5WS)*
* Subject has signed institutional review board (IRB)-approved informed consent form

Exclusion Criteria:

* Subject takes any medication or dietary supplement regularly that affects blood clotting (e.g., Coumadin, aspirin, clopidogrel) or increases the risk of bleeding/bruising
* Subject has had prior surgery that alters the subcutaneous anatomy of the target treatment sites
* The investigator is unable to substantially lessen facial lines by physical separation
* Subject has undergone another facial cosmetic procedures at or above the level of the cheekbones within the past 6 months
* Subject is participating in another facial cosmetic research study

Patient has any of following conditions:

* History of facial nerve palsy
* Marked facial asymmetry
* Ptosis
* Excessive dermatochalasis
* Deep dermal scarring
* Thick sebaceous skin
* History of neuromuscular disorder
* Chronic dry eye symptoms
* Allergy or intolerance to lidocaine
* Other local skin condition (eg, skin infection) at target treatment site
* Any physical or psychiatric condition that in the investigator's opinion would prevent adequate study participation

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Wrinkle Severity and incidence of device-related serious adverse events | Up to 4 months
  * Effectiveness endpoint: Wrinkle severity in the target area in animation at 30 days post-treatment as rated by the investigator using the 5-point grading scale.
  * Safety endpoint: Incidence of device-related serious adverse events (DSAE).

SECONDARY OUTCOMES:
Wrinkle Severity | Up to 4 months
  • Investigators' rating of wrinkle severity in the target area in animation immediately post-treatment, at 1 and 7 days post-treatment and at 30-day intervals for 120 days after treatment
Independent Assessment | Up to 4 months
  • Independent reviewers' ratings of forehead wrinkle severity at rest and in animation at 30-days post-treatment
Global assessment | Up to 4 months
  • Subjects' global assessment of change in appearance of target area immediately post-treatment, at 1 and 7 days post-treatment and at 30-day intervals for 120 days after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Aesthetics Research Center, Redwood City, California, United States